CLINICAL TRIAL: NCT07202247
Title: A Phase II Randomized Study of Interventions for Metabolic Protection Against Cardiometabolic Toxicity During Androgen Deprivation Therapy (IMPACT-ADT)
Brief Title: Metabolic Interventions (Time-Restricted Eating, GLP1 Receptor Agonist, and Heart Healthy Diet) to Improve Cardiometabolic Health in Prostate Cancer Patients During Androgen Deprivation Therapy, IMPACT-ADT Trial
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 25332; NCI-2025-06197 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 25332 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2025-09-18; First posted 2025-10-01 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Prostate Carcinoma; Recurrent Prostate Carcinoma
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Androgen Antagonists; Behavior Therapy; Specimen Handling; Radiotherapy; Radiation; Referral and Consultation; semaglutide; Tirzepatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm 1 (TRE) (Experimental): Patients receive RT and ADT per SOC, as well as participate in an overnight fast over 16 hours on at least 5 days weekly for 6 months. Patients also receive TRE reminders, dietary education, and complete survey and food diary collection via the Oncpatient Companion Mobile app. In addition, patients receive diet/lifestyle counseling as per AHA HHD guidelines and AHA Life Essential 8 recommendations with personalized caloric intake for 6 months. Patients may may optionally wear an activity tracker throughout the trial. Additionally, patients undergo CT, blood sample collection throughout the study and may optionally undergo a coronary computerized tomography angiography throughout the study.
  Interventions: Drug: Antiandrogen Therapy; Behavioral: Behavioral Intervention; Procedure: Biospecimen Collection; Procedure: Cardiac Computerized Tomographic Angiography; Procedure: Computed Tomography; Other: Electronic Health Record Review; Other: Internet-Based Intervention; Behavioral: Lifestyle Counseling; Other: Medical Device Usage and Evaluation; Other: Nutritional Intervention; Other: Questionnaire Administration; Radiation: Radiation Therapy; Other: Short-Term Fasting
- Arm 2 (semaglutide, tirzepatide) (Experimental): Patients receive RT and ADT per SOC for 6 months. Patients receive a referral to an endocrinologist and receive semaglutide or tirzepatide SC QW for 6 months in the absence of disease progression or unacceptable toxicity. Patients also receive dietary education and complete survey and food diary collection via the Oncpatient Companion Mobile app. In addition, patients receive diet/lifestyle counseling as per AHA HHD guidelines and AHA Life Essential 8 recommendations with personalized caloric intake for 6 months. Patients may may optionally wear an activity tracker throughout the trial. Additionally, patients undergo CT, blood sample collection throughout the study and may optionally undergo a coronary computerized tomography angiography throughout the study.
  Interventions: Drug: Antiandrogen Therapy; Procedure: Biospecimen Collection; Procedure: Cardiac Computerized Tomographic Angiography; Procedure: Computed Tomography; Other: Electronic Health Record Review; Other: Internet-Based Intervention; Behavioral: Lifestyle Counseling; Other: Medical Device Usage and Evaluation; Other: Nutritional Intervention; Other: Questionnaire Administration; Radiation: Radiation Therapy; Other: Referral; Drug: Semaglutide; Drug: Tirzepatide
- Arm 3 (AHA HDD) (Active Comparator): Patients receive RT and ADT per SOC for 6 months. Patients receive diet/lifestyle counseling as per AHA HHD guidelines and AHA Life Essential 8 recommendations with personalized caloric intake for 6 months. Patients also receive dietary education and complete survey and food diary collection via the Oncpatient Companion Mobile app. Patients may may optionally wear an activity tracker throughout the trial. Additionally, patients undergo CT, blood sample collection throughout the study and may optionally undergo a coronary computerized tomography angiography throughout the study.
  Interventions: Drug: Antiandrogen Therapy; Procedure: Biospecimen Collection; Procedure: Cardiac Computerized Tomographic Angiography; Procedure: Computed Tomography; Other: Electronic Health Record Review; Other: Internet-Based Intervention; Behavioral: Lifestyle Counseling; Other: Medical Device Usage and Evaluation; Other: Nutritional Intervention; Other: Questionnaire Administration; Radiation: Radiation Therapy

INTERVENTIONS:
Drug: Antiandrogen Therapy — Given ADT
  Other Names: ADT; Androgen Deprivation Therapy; Androgen Deprivation Therapy (ADT); Anti-androgen Therapy; Anti-androgen Treatment; Antiandrogen Treatment; Hormone Deprivation Therapy; Hormone-Deprivation Therapy
Behavioral: Behavioral Intervention — Receive fasting reminders via Oncpatient Companion Mobile Application
  Other Names: Behavior Conditioning Therapy; Behavior Modification; Behavior or Life Style Modifications; Behavior Therapy; Behavioral; Behavioral Interventions; Behavioral Modification; Behavioral Therapy; Behavioral Treatment; Behavioral Treatments
  Arms: Arm 1 (TRE)
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Cardiac Computerized Tomographic Angiography — Undergo a coronary computerized tomography angiography
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Other: Electronic Health Record Review — Ancillary studies
Other: Internet-Based Intervention — Complete survey and food diary collection via Oncpatient Companion Mobile Application
Behavioral: Lifestyle Counseling — Receive diet and lifestyle counseling
Other: Medical Device Usage and Evaluation — Wear an activity tracker
Other: Nutritional Intervention — Receive AHA HHD guidelines
Other: Nutritional Intervention — Receive AHA Life Essential 8 recommendations with personalized caloric intake
Other: Questionnaire Administration — Ancillary studies
Radiation: Radiation Therapy — Undergo RT
  Other Names: Cancer Radiotherapy; Energy Type; ENERGY_TYPE; Irradiate; Irradiated; Irradiation; Radiation; Radiation Therapy, NOS; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation
Other: Referral — Receive a referral to an endocrinologist
  Other Names: Referred
  Arms: Arm 2 (semaglutide, tirzepatide)
Drug: Semaglutide — Given SC
  Other Names: Ozempic; Rybelsus; Wegovy
  Arms: Arm 2 (semaglutide, tirzepatide)
Other: Short-Term Fasting — Participate in an overnight fast
  Other Names: Intermittent Fasting; Short-term Intermittent Fasting
  Arms: Arm 1 (TRE)
Drug: Tirzepatide — Given SC
  Arms: Arm 2 (semaglutide, tirzepatide)

SUMMARY:
This phase II trial compares the effect of time-restricted eating (TRE) and glucagon-like peptide-1 (GLP1) receptor agonists (RA), semaglutide and tirzepatide, to an American Heart Association (AHA) heart healthy diet (HHD) intervention on heart and blood vessel health (cardiovascular system) and how the body processes food for energy (metabolic system) in prostate cancer patients undergoing androgen deprivation therapy (ADT). Prostate cancer patients who are receiving hormonal therapy (ADT) are at an increased risk of cardiovascular disease. This is thought to be due to treatment-related metabolic changes which may result in increased weight, body fat, insulin resistance and an increased risk of heart attack, stroke or other heart and blood vessel problems. TRE (also known as intermittent fasting) is an eating plan that alternates between fasting and non-fasting periods. This approach limits calorie intake to a specific window of time each day. GLP1-RAs, semaglutide and tirzepatide are in a class of medications called incretin mimetics. They work by helping the pancreas to release the right amount of insulin when blood sugar levels are high. Insulin helps move sugar from the blood into other body tissues where it is used for energy. They also slow the movement of food through the stomach and may decrease appetite and cause weight loss. The AHA HHD guidelines may be an effective method to help people learn about following a heart healthy eating plan. This may lower their risk of cardiovascular disease. Metabolic interventions, TRE and GLP1-RA, may be more effective than an AHA HHD intervention alone in improving cardiovascular and metabolic health in prostate cancer patients undergoing ADT.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Evaluate whether metabolic interventions, including TRE and GLP1-RA treatment, improve the cardiometabolic health of prostate cancer (PCa) patients undergoing ADT.

SECONDARY OBJECTIVES:

I. Characterize the metabolic and inflammatory profiles for patients at high risk of ADT-associated cardiometabolic disease during ADT.

II. Evaluate tolerability and feasibility of concurrently using GLP1-RA or performing TRE during short-term ADT.

III. Examine if metabolic interventions, including TRE and GLP1 RA treatment, are associated with improved patient quality of life.

EXPLORATORY OBJECTIVES:

I. Define the impact of metabolic interventions, including TRE and GLP1 RA treatment, on ADT-induced metabolome-inflammasome dysfunction.

II. Evaluate the impact of metabolic interventions, including TRE and GLP1 RA treatment, on clonal dynamics following ADT.

III. Evaluate how metabolic interventions, including TRE and GLP1 RA treatment, impact coronary plaque characteristics in PCa patients undergoing ADT.

OUTLINE: Patients are randomized to 1 of 3 arms.

ARM 1 (TRE): Patients receive radiation therapy (RT) and ADT per standard of care (SOC), as well as participate in an overnight fast over 16 hours on at least 5 days weekly for 6 months. Patients also receive TRE reminders, dietary education, and complete survey and food diary collection via the Oncpatient Companion Mobile Application (app). In addition, patients receive diet/lifestyle counseling as per AHA HHD guidelines and AHA Life Essential 8 recommendations with personalized caloric intake for 6 months. Patients may may optionally wear an activity tracker throughout the trial.

ARM 2 (GLP1-RA): Patients receive RT and ADT per SOC for 6 months. Patients receive a referral to an endocrinologist and receive semaglutide or tirzepatide subcutaneously (SC) once weekly (QW) for 6 months in the absence of disease progression or unacceptable toxicity. Patients also receive dietary education and complete survey and food diary collection via the Oncpatient Companion Mobile app. In addition, patients receive diet/lifestyle counseling as per AHA HHD guidelines and AHA Life Essential 8 recommendations with personalized caloric intake for 6 months. Patients may may optionally wear an activity tracker throughout the trial.

ARM 3 (AHA HHD): Patients receive RT and ADT per SOC for 6 months. Patients receive diet/lifestyle counseling as per AHA HHD guidelines and AHA Life Essential 8 recommendations with personalized caloric intake for 6 months. Patients also receive dietary education and complete survey and food diary collection via the Oncpatient Companion Mobile app. Patients may may optionally wear an activity tracker throughout the trial.

Additionally, patients undergo computed tomography (CT), blood sample collection throughout the study, and may optionally undergo a coronary computerized tomography angiography throughout the study.

After completion of study intervention, patients are followed up at 30 days and at 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Documented informed consent of the participant
* English, Spanish or Mandarin-speaking
* Agreement to allow the use of archival tissue from diagnostic tumor biopsies

  * If unavailable, exceptions may be granted with study principal investigator (PI) approval
* Male
* Aged: 30-79
* Eastern Cooperative Oncology Group (ECOG) 0-2
* High burden of cardiovascular comorbidities who would be eligible for insurance coverage for GLP1-RA therapy defined as:

  * Body mass index (BMI) of ≥ 30 kg/m^2 or
  * BMI ≥ 27 kg/m^2 in the presence of at least one weight-related comorbid condition (e.g. hypertension, type 2 diabetes mellitus, dyslipidemia)
* Prostate cancer defined as one of the following:

  * National Comprehensive Cancer Network (NCCN) intermediate risk prostate cancer receiving definitive radiation with a plan to undergo ADT for 6 months
  * Biochemical persistent or recurrent prostate cancer status post prostatectomy receiving salvage radiation with a plan to undergo ADT for 6 months

Exclusion Criteria:

* Currently engaging in strict macronutrient/time limited diet, including ketogenic, low-carb, paleo, or warrior diet
* Currently under GLP1-RA therapy
* Poorly controlled diabetes
* Unable to undergo time-restricted diet
* Contraindications for GLP1-RA therapy: including hypersensitivity to the drug, personal history of pancreatitis, personal or family history of medullary thyroid cancer or multiple endocrine neoplasia syndrome type 2, end-stage renal disease
* Other active disease deemed not eligible to participant in the study according to treating physician
* Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics)

Ages: 30 Years to 79 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-01-23 (Actual); Primary Completion 2028-04-09 (Estimated); Study Completion 2028-04-09 (Estimated)

PRIMARY OUTCOMES:
Changes in the 10-year risk of cardiovascular disease | At completion of 6 months of androgen deprivation therapy (ADT) and at 12 months follow up after completion of ADT
  The changes in the American Heart Association Predicting Risk of cardiovascular disease (CVD) EVENTs (AHA PREVENT) risk score will be compared between glucagon-like peptide-1 receptor agonist (GLP1-RA) versus (vs.) AHA heart healthy diet (AHA HHD) interventions using a 2-group t-test with a 0.050 one-sided significance level.
Changes in the 10-year risk of cardiovascular disease | At completion of 6 months of ADT and at 12 months follow up after completion of ADT
  The changes in the AHA PREVENT risk score will be compared between time-restricted eating (TRE) vs. AHA HHD interventions using a 2-group t-test with a 0.050 one-sided significance level.

SECONDARY OUTCOMES:
Changes in the 10-year risk of cardiovascular disease | At completion of 6 months of ADT and at 12 months follow up after completion of ADT
  The changes in the AHA PREVENT risk score will be compared between GLP1-RA vs. TRE interventions.
Incidence of de novo metabolic syndrome | At completion of 6 months of ADT and at 12 months follow up after completion of ADT
Changes in visceral adiposity | At completion of 6 months of ADT and at 12 months follow up after completion of ADT
  Will be measured using computed tomography and bioelectrical impedance analysis.
Changes in muscle mass | At completion of 6 months of ADT and at 12 months follow up after completion of ADT
  Will be measured using computed tomography and bioelectrical impedance analysis.
Evidence of endothelial dysfunction | At completion of 6 months of ADT and at 12 months follow up after completion of ADT
  Will be measured by flow mediated dilation of the brachial artery.
Percent of patients who successfully complete interventions | Up to 12 months after completion of ADT
  Tolerability and feasibility will be defined as at least 70% of enrolled patients successfully completing the interventions for a minimum of 70% of the study duration.
Quality of life - International Prognostic Scoring System | At baseline and up to 12 months after completion of ADT
  Will be measured using the International Prognostic Scoring System.
Quality of life - Sexual Health Inventory for Men | At baseline and up to 12 months after completion of ADT
  Will be measured using the Sexual Health Inventory for Men.
Quality of life - Merrick rectal function | At baseline and up to 12 months after completion of ADT
  Will be measured using the Merrick rectal function.
Quality of life - Patient Reported Outcomes Measurement Information System 29 | At baseline and up to 12 months after completion of ADT
  Will be measured using the Patient Reported Outcomes Measurement Information System 29.

CONTACTS AND LOCATIONS:
Overall Officials: Rose Li, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States